CLINICAL TRIAL: NCT05040165
Title: Investigation on Failure Time Analysis of a New TPE Material in the Iceform Liner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CIP2019052102
Record Dates: First submitted 2020-11-18; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Prosthesis Failure
MeSH Terms: conditions — Prosthesis Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Failure time analysis (Experimental): The primary objective is to evaluate the durability of the investigational device over its intended use lifetime (i.e. warranty period), specifically relating to any defect in the TPE material. Additionally, to gather information on the rate of side-effects, i.e. skin rashes, sores, etc.
  Secondary objectives relate to gather information on how amputees use the liner, specifically:
  * Intensity of use (days/week and hours/day)
  * Alternation; i.e. switching every other day between liners
  * Use of personal hygiene or cosmetic products
  The following performance and safety aspects are to be verified:
  • The ICEFORM line of devices are durable over their intended use lifetime.
  Interventions: Device: Iceform liner and sleeve

INTERVENTIONS:
Device: Iceform liner and sleeve — Subjects will be asked to use the investigational device as their primary prosthesis for up to 6 months. TPE material durability evaluated through monthly online questionnaires.

SUMMARY:
Durability evaluation of a new material blend in the Iceform liner and Iceform sleeve.

DETAILED DESCRIPTION:
Potential subjects will be identified from the customer base of a relevant clinic. If a potential participant may fit the inclusion and exclusion criteria, he/she will be contacted by a Co-Investigator (CI) via telephone. During the telephone call the CI will verify if they are interested in participating in a study and will initiate the enrollment procedure. If interest is expressed at this point they will answer some screening questions and if the eligibility criteria is met the subject is offered to enroll by getting a study invite through ProofPilot, the EDS, and an appointment to come in for initial fitting will be set up. Questions relating to the duration of the study, number of clinical visits required, and the investigational device will be answered at this time.

Following this the subject will log into ProofPilot online and go through the e-ICF, if signed, the subject will answer a profile questionnaire.

The next step will be an appointment, subject comes into their clinic and gets the investigational device. In some cases, the subject will get the liner shipped to their home address. This will only be done upon subjects request due to long distance from clinic. And only for very confident prosthetic users which are used to handle a new liner by themselves.

Potential risk of participating in the investigation will be explained to the subject at this point. The CIs will communicate to the study monitors the number of users that have been identified that meet the inclusion/exclusion criteria and are willing to participate.

During the clinical visit the subjects will only be fitted to the Iceform investigational liner. Profile and relevant contact information will already have been collected via the EDS.

Subjects will then receive a prompt monthly, either via email, SMS or smartphone notification, to fill in the EDS questionnaire, and perform any tasks as applicable. If a subject reports a failure he/she will be instructed to stop using the liner, the remaining gift cards will be delivered and their participation ends. Otherwise, participation will end at 6 months.

The subject gets to keep the investigational device at the end of the study, therefore there is no need for an additional visit.

Subjects that report a failure of the TPE material may be contacted by the Coordinating Investigator or CI if the root cause of the failure cannot be confidently determined from the data collected with the EDS system.

ELIGIBILITY:
Inclusion Criteria:

* Trans-tibial amputee
* Uses an Iceform or Willow Wood Alpha Classic (Uniform profile) liner
* Willing and able to participate in the study and follow the protocol
* Confident prosthetic users for more than 3 months
* Older than 18 years

Exclusion Criteria:

* Participating in another research study
* Participants of another research study during previous 2 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-12-08 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Cumulative failure rate | 3 months
  TPE material durability
Cumulative failure rate | 6 months
  TPE material durability

CONTACTS AND LOCATIONS:
Overall Officials: Justin L Pratt, CP, Principal Investigator — Össur
Locations (1):
- ProofPilot, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No